CLINICAL TRIAL: NCT04098237
Title: Pancreatic-enzyme Replacement Therapy With Pancreaze (Pancrelipase) Delayed-release in Addition to Standard of Care for Borderline Resectable, Locally Advanced, and Advanced Pancreatic Adenocarcinoma Patients (PANCAX-3) With Cachexia and Exocrine Pancreatic Insufficiency
Brief Title: Pancreaze (Pancrelipase) for Patients With Pancreatic Adenocarcinoma With Cachexia and Exocrine Pancreatic Insufficiency
Acronym: PANCAX-3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew Hendifar, MD (Other)
Collaborators: VIVUS LLC (Industry)
Responsible Party: Sponsor-Investigator, Andrew Hendifar, MD, Sponsor-Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2018-29-HENDIFAR-PNCX3
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard of care treatment with Pancreaze (pancrelipase) (Experimental): Pancrelipase capsules; 84,000 IU lipase units per main meal and 42,000 IU lipase units per snack; for 24 weeks
  Interventions: Drug: Pancrelipase

INTERVENTIONS:
Drug: Pancrelipase — Pancrelipase delayed-release capsules

SUMMARY:
The objective of this study is to assess weight stability, functional changes, and quality of life when Pancreaze (pancrelipase) delayed-release 84,000-lipase units (capsules), for main meals, and 42,000-lipase units (capsules), for snacks, are added to standard of care in patients with exocrine pancreatic insufficiency due to pancreatic adenocarcinoma. This will be the first prospective study of this particular formulation in addition to standard of care in advanced pancreatic cancer patients. We will treat 40 consecutive patients with borderline resectable, locally advanced and advanced pancreatic cancer patients who present with weight loss and exocrine pancreatic insufficiency with this advanced formulation of Pancreaze.

ELIGIBILITY:
Inclusion Criteria:

1. Borderline resectable, locally advanced, and advanced pancreatic cancer patients (can include new or recurrent diagnosis) referred to SOCCI-CSMC (Samuel Oschin Cancer Center - Cedars Sinai Medical Center)
2. Age ≥ 18 years.
3. ECOG performance status 0-1 or Karnofsky PS >60%
4. Clinical diagnosis of exocrine pancreatic insufficiency
5. Cachexia defined as at least 5% weight loss in the presence of chronic illness, within any 6-month period prior to screening OR as documented by the medical physician based on standard diagnosis of cachexia
6. Life expectancy of greater than 3 months, in the opinion of the investigator.
7. Patients must have normal organ and marrow function as defined below:

   * Absolute Neutrophil Count (ANC) ≥ 500/mcL
   * Platelets ≥ 50,000/mcL
   * Total bilirubin ≤ 5X upper limit of normal (ULN)
   * AST(SGOT)/ALT(SGPT) ≤ 5 X ULN
   * Creatinine OR creatinine clearance ≤ 3 times the upper limit of normal OR ≥ 30 mL/min/1.73 m² for patients with creatinine levels above normal.
   * Note: Patients with biliary stents are eligible provided that all other inclusion criteria are met.
8. Woman of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the time of signing the informed consent form, for the duration of study participation, and for at least 30 days after discontinuing from study treatment.
9. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Women who are pregnant or are breastfeeding
3. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
4. Unable to swallow intact capsules
5. Fibrosing colonopathy: Patients with history of fibrosing colonopathy have been reported to experience advancement to colonic strictures with doses of lipase>6000 units/kg/meal over prolonged periods of time.
6. History of chronic illness associated with malabsorption or nutrient deficiency including but not limited to chronic pancreatitis, cystic fibrosis, celiac disease, Crohn's disease, pernicious anemia and/or prior intestinal resection.
7. Coexistent other primary malignancy
8. Pregnancy, breastfeeding, or of childbearing potential and not willing to use methods of birth control during the study
9. Active drug abuse or intoxication with any substance including alcohol (blood alcohol content >0.08%, legal driving limit)
10. Known allergy to any of the active ingredients in pancreatic enzyme supplementation
11. Concurrent use of pancreatic enzyme supplementation or over the counter supplements which contain lipase, protease, and amylase as active ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2027-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hendifar, MD, MPH, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Started | 36
Completed | 30
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Median Age and Inter-Quartile Range for all evaluable participants
  years | 70 [52 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Completing Pancreatic Enzyme Replacement Therapy During the First 8 Weeks of the Study: Daily Compliance Diary
Description: Adherence to therapy of at least 50% of the needed total lipase units, recorded using a daily compliance diary.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 30
Participants | 29

2. Secondary Outcome: Mean Change in Weight From Baseline Through the End-of-study Visit
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 29
lbs | -2.1931 (6.163831)

3. Secondary Outcome: Mean Change in Calories Consumed From Baseline Through the End-of-study Visit
Description: As measured by Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool. The ASA24 is a system to collect 24-hour food recalls and provide complete nutrient analysis of the foods and beverages consumed during the collection timeframe. The tool is used in this study to measure total calories consumed.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: calories
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 27
calories | -169.2075 (969.6394)

4. Secondary Outcome: Mean Change in Stool Frequency From Baseline Through Cycle 3 Day 1
Description: As measured by patient reported number of bowel movements in the past 24 hours. In this study, higher numbers represent more severe symptoms; a reduction in number of bowel movements in the past 24 hours represents improvement in symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: bowel movements/day
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 27
bowel movements/day | -0.96296 (2.457038)

5. Secondary Outcome: Mean Change in Stool Consistency From Baseline Through Cycle 3 Day 1
Description: As measured by patient reported stool consistency using the Bristol Stool Chart.The Bristol Stool Chart is a diagnostic scale to classify stool into 7 different groups, ranging from Type 1-7 (indicating solid to liquid consistency or time spent longest in the bowel to least time in the bowel). A normal stool should be either Type 3 or Type 4 (middle of the scale). Worsening of stool consistency is denoted by classifications located closer to the extreme ends of the scale (Type 1 or Type 7).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on Bristol Stool Form Scale
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 27
units on Bristol Stool Form Scale | -0.407407 (1.906654)

6. Secondary Outcome: Mean Change in Serum Levels of Fat-soluble Vitamins From Baseline - Vitamin A
Time Frame: 6 months
Population: Some patients were missing vitamin values.
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 30
mcg/dL | -0.5 (14.70231)

7. Secondary Outcome: Mean Change in Serum Levels of Fat-soluble Vitamins From Baseline - Vitamin D
Time Frame: 6 months
Population: Some patients were missing vitamin values
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 21
ng/mL | -5.37619 (12.44841)

8. Secondary Outcome: Mean Change in Serum Levels of Fat-soluble Vitamins From Baseline - Vitamin E
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 20
mg/L | 0.495 (3.988863)

9. Secondary Outcome: Mean Change in Serum Levels of Fat-soluble Vitamins From Baseline - Vitamin K
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 17
pg/mL | -27.47059 (676.6716)

10. Secondary Outcome: Mean Change in Serum Levels of Fat-soluble Vitamins From Baseline - Vitamin K PT
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 21
pg/mL | -0.2190476 (2.82889)

11. Secondary Outcome: Change in Microbiome From Baseline
Description: Microbiome analysis of stool samples
Time Frame: 8 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Mean Change in Daily Activity (Steps Taken) From Baseline
Description: As measured by continuous daily wearable activity monitor
Time Frame: 6 months
Measure: Mean (Standard Error); unit: steps/day
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 30
steps/day | -0.3 (3.8)

13. Secondary Outcome: Mean Change in Daily Activity (Stairs Climbed) From Baseline
Description: As measured by continuous daily wearable activity monitor
Time Frame: 6 months
Measure: Mean (Standard Error); unit: stair steps/day
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 30
stair steps/day | 1332.6 (539.4)

14. Secondary Outcome: Mean Change in Sleep Disturbance From Baseline
Description: As measured by continuous daily wearable activity monitor
Time Frame: 6 months
Measure: Mean (Standard Error); unit: hours/night
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 30
hours/night | 0.5 (0.83)

15. Secondary Outcome: Mean Change in Duration of Sleep Disturbances From Baseline
Description: As measured by continuous daily wearable activity monitor. An absolute change in the percentage of time during nighttime sleep in which participants experienced sleep disturbance is being reported.An absolute change in percent is understood to be calculated as the value at the later time point minus the value at the earlier time point (e.g., value at 6 months minus value at baseline).
Time Frame: 6 months
Measure: Mean (Standard Error); unit: % of nighttime sleep
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 30
% of nighttime sleep | 4.43 (1.3)

16. Secondary Outcome: Mean Change in Average Heart Rate From Baseline
Description: As measured by continuous daily wearable activity monitor
Time Frame: 6 months
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 30
beats per minute | 0.8 (2.6)

17. Secondary Outcome: Mean Change in Peak Heart Rate From Baseline
Description: As measured by continuous daily wearable activity monitor
Time Frame: 6 months
Measure: Mean (Standard Error); unit: BPM
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 30
BPM | 9.6 (5.4)

18. Secondary Outcome: Mean Change in Daily Active Minutes From Baseline
Description: As measured by continuous daily wearable activity monitor
Time Frame: 6 months
Measure: Mean (Standard Error); unit: minutes/day
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
Number analyzed (Participants) | 30
minutes/day | 3.0 (6.7)

ADVERSE EVENTS:
Time Frame: 6 months
Description: The investigator or designee is responsible for ensuring that adverse events (both serious and non-serious) observed by the clinical team or reported by the subject which occur after the subject has initiated treatment and until the 30-day end-of-study visit, are fully recorded in the subject's medical records Adverse events will be assessed from time of treatment initiation for the duration of the study treatment period until the end-of-study visit.
Arm/Group | Standard of Care Treatment With Pancreaze (Pancrelipase)
All-Cause Mortality (participants affected / at risk) | 21/30
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 7/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Treatment With Pancreaze (Pancrelipase) (N=30)
Ascites (General disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Biliary Tract Infection (Infections and infestations) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1)
Colotis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Hepatic Infection (Infections and infestations) | 1 (1)
Hepatic Infection (Hepatobiliary disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Other (General disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (2)
Sepsis (General disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Urinary Tract Infections (Infections and infestations) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Visceral Arterial Ischemia (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Treatment With Pancreaze (Pancrelipase) (N=30)
Abnominal Pain (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT04098237/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT04098237/ICF_001.pdf